CLINICAL TRIAL: NCT04291261
Title: Phase II Multicenter Study of Extracorporal Photopheresis With UVADEX Plus Standard Steroid Treatment for High Risk Acute Graft-versus-host Disease
Brief Title: Extracorporal Photopheresis With UVADEX Plus Standard Steroid Treatment for High Risk Acute Graft-versus-host Disease
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Universitätsklinikum Hamburg-Eppendorf (Other)
Collaborators: Therakos (Industry); University Medical Center Regensburg (Unknown); Arbeitskreis Klinische Forschung PD Dr. med. Seiler GmbH (Network)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MAGIC-HR-ECP
Record Dates: First submitted 2020-02-19; First posted 2020-03-02 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: Acute-graft-versus-host Disease
Keywords: Acute-graft-versus-host Disease; Allogeneic Stem Cell Transplantation; Ann Arbor GvHD Scoring
MeSH Terms: interventions — Methoxsalen

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Extracorporeal photopheresis (ECP) with Uvadex (Other): Patients in this single Arm study all receive the intervention consisting of ECP with Uvadex plus the standard of care treatment which consists of systemic corticosteroids 2mg/kg. Response to treatment will be evaluated on day 28. Patients will receive study treatment till day 56 and thereafter be followed until 1 year.
  Interventions: Drug: Uvadex

INTERVENTIONS:
Drug: Uvadex — Extracorporeal photopheresis (ECP) with Uvadex is scheduled 3x/week in weeks 1+2, 2x/week thereafter till day 28 and 1x/week till day 56

SUMMARY:
This is a single arm phase 2 trial which includes patients with high risk acute GVHD defined as Ann Arbor score 2 or 3. The purpose of the study is to improve the outcome of these patients in terms of response to treatment and treatment related mortality. All patients will receive the study intervention (ECP with Uvadex). The study hypothesis is that the treatment plan will produce a day 28 complete response rate higher than or equal to 52%, which will represent an improvement of 15% compared with the standard of care (37%). The rate of complete response to standard of care treatment is based on observed data in similar patients treated within the Mount Sanai Acute GVHD International Consorium (MAGIC). Patients will be treated for 56 days and followed for one year to also enable evaluation of long term outcome.

DETAILED DESCRIPTION:
This study is a single arm phase 2 study for adult patients who have acute GVHD Grade II-IV according to Glucksberg and Ann Arbor score 2 or 3 after first allogeneic stem cell transplantation. The staging according to Glucksberg is based on clinical parameters while Ann Arbor scoring is based on the MAGIC biomarkers. Patients will receive standard acute GVHD treatment consisting of 2mg/kg methylprednisolone plus extracorporeal photopheresis (ECP) with Uvadex. Day 0 of the study will be the first day of ECP, which will be performed 3x weekly for the first 2 weeks, 2x weekly for the next two weeks and thereafter once weekly until day 56. A taper schema for methylprednisolone is proposed but not obligatory. Patients will be followed until one year after start of ECP.

The study plans to enroll 72 patients in order to be able to detect a 15% difference in rate of complete responses on day 28, assuming a type I error rate of 0.05. Patients treated on this study will have three possible comparators:

* Cohort of patients with high risk aGvHD who received standard treatment and whose data were prospectively reported to MAGIC during the last 2 years preceding the trial
* Cohort of patients with high risk aGvHD who received standard treatment and whose data are reported to MAGIC during the trial period
* Cohort of patients with high risk aGvHD treated within the ongoing prospective MAGIC USA phase 2 Trial

Treatment:

Prior to an ECP treatment each patient will be assessed by a physician to verify that the patient is acceptable for ECP treatment. This assessment will include vital signs (diastolic and systolic blood pressures, pulse, temperature) which will be taken prior to and at the end of each ECP treatment. Blood cell counts will be analyzed prior to each treatment. If a patient's WBC count is below 1 X 109/L or platelet count is below 20 X 109/L ECP should be postponed until rise in WBC or platelet counts. Platelet transfusions and use of cytokines is permitted. Whenever possible, peripheral venous access is preferable to central venous catheters. In patients with platelet counts below 40 X 109/L acid citrate dextrose (ACD) instead of heparin should be used for ECP. When severe acute infections occur during study ECP should be discontinued until the infection has been controlled under appropriate therapy

Topical therapy for acute GvHD of the skin and non-absorbable steroids for GI GvHD are allowed. Ancillary/supportive care measures for acute GvHD such as the use of anti-motility agents for diarrhea, including octreotide, is allowed at the discretion of the treating physician. Use of ursodiol to prevent/reduce gall bladder sludging, or prevent hepatic transplant complications is also allowed according to institutional guidelines.

In addition to prescribed study drug plus corticosteroids, all patients should receive the following:

* Transfusion support per institutional practice
* Anti-infective prophylaxis against herpes virus is required but otherwise institutional practice can be followed for the medication to be used and the dosing
* Anti-infective prophylaxis against Pneumocystis jiroveci, bacterial and fungal infections according to standard institutional guidelines.
* Anti-infective prophylaxis against fungi (aspergillosis) is required but otherwise institutional practice can be followed
* Pre-emptive monitoring and treatment for CMV and EBV infections are required but otherwise institutional practice can be followed.

Efficacy and stopping rules:

Efficacy of the treatment plan will be assessed by the proportion of patients with complete response at day 28. The treatment plan will be considered efficacious if it produces a day 28 CR rate of ≥ 52%, representing an improvement over the day 28 CR rate of approximately 15% achieved with the standard of care. Stopping boundaries for efficacy are presented in Table 5, in terms of the number of observed positive responses out of the total number observed. Our expectation is represented by a prior distribution for a positive response that has a mean of 0.37, or 37%. Characterizing our expectation as a distribution of values, rather than a fixed value, naturally accounts for uncertainty in the response. The prior is based on observed data treating similar patients with the standard of care. More specifically, let θS be the day 28 CR rate of patients treated with the standard of care. Likewise, let θE be the day 28 CR of patients treated with ECP and high dose systemic corticosteroid. Assume that θS ~ beta (37, 63) and θE ~ beta (0.74, 1.26) so that each prior has a mean of 0.37. Let the improvement of the experimental treatment over the standard, δ, be 0.1. The study will be stopped when P (θS + δ >θE |observed data)>0.90.

The boundaries provide guidelines for determining when treatment with ECP and high dose systemic corticosteroid is inferior to what would be expected if patients were treated with the standard of care. We will initiate these guidelines with the 10th outcome, and enroll a maximum of 72 patients.

Further stopping rules:

For the individual patient:

Any of the following criteria will lead to study discontinuation:

* Inter-current illness that prevents further administration of treatment
* Unacceptable adverse event(s)
* Patient voluntarily withdraws from treatment OR
* General or specific changes in the patient's condition render the patient unacceptable for further treatment in the judgment of the investigator or Sponsor

The reason for ending protocol therapy and the date the patient was removed from treatment will be documented in the study record. All patients who discontinue treatment should comply with protocol specific follow-up procedures as outlined in Section 13.13. The only exception to this requirement is when a patient withdraws consent for all study procedures.

Patients may withdraw from the study treatment at their request at any time. If they withdraw, they will be asked to perform a study termination visit and be documented in eCRF as "early termination". The reasons should be documented in the eCRF.

For the entire study cohort:

The whole study can be discontinued by the Coordinating Investigator in case of excessive toxicity.

For safety reasons, a study termination visit should be performed and the included patients should be further followed-up until disease progression or death from any cause (relapse or other reason).

Once we have enrolled 10 patients, and for additional patients thereafter, we will assess the cumulative number of patients with overall response and NRM and stop the trial if the observed number responses or NRM equals or exceeds the thresholds specified in section 19.

ELIGIBILITY:
Inclusion Criteria:

1. New onset high risk acute GvHD (Ann Arbor score 2/3 as defined in Appendix A) following allogeneic SCT. Any clinical severity in accordance with Glucksberg grade II-IV is eligible.
2. Any donor type (e.g., related, unrelated) or stem cell source (bone marrow, peripheral blood, cord blood). Recipients of non-myeloablative and myeloablative transplants are eligible.
3. No prior systemic treatment for acute GvHD except for a maximum of 7 days of methylprednisolone ≤2 mg/kg/day (or IV methylprednisolone equivalent) during the period from initiation of systemic steroid treatment for acute GvHD until study therapy begins. Topical skin steroid treatment and non-absorbable oral steroid treatment for GI GvHD are permissible.
4. Age 18 years or older.
5. Platelet count > 25.000 (including platelet support)
6. Eastern Coorperative Oncology Group (ECOG) score of 0≤2 unless due to aGvHD
7. Negative pregnancy test within 10 days before start of study if the patient is a woman of child-bearing Age
8. Direct bilirubin must be <2 mg/dL unless the elevation is known to be due to Gilbert syndrome or aGvHD within 3 days before screening.
9. ALT/SGPT and AST/SGOT must be <5 x the upper limit of the normal range within 3 days before screening.
10. Females/Males who agree to comply with the applicable contraceptive requirements of the protocol.
11. Written informed consent from patient.
12. Biopsy of acute GvHD target organ is strongly recommended but not required. Enrollment should not be delayed for biopsy or pathology results. Patients who do not enroll within 5 working days of Initiation of systemic steroid treatment for acute GvHD are not permitted to participate

Exclusion Criteria:

1. Progressive or relapsed malignancy
2. Uncontrolled active infection
3. Patients with chronic GvHD
4. History of or current diagnosis of progressive multifocal leukoencephalopathy (PML)
5. Pregnant or nursing (lactating) women
6. Use of other drugs for the treatment of acute GvHD apart from ongoing GvHD prophylaxis and corticosteroids
7. Patients on dialysis
8. Patients requiring ventilator support
9. Evidence of known infection with human immunodeficiency virus (HIV) or active hepatitis B
10. Investigational agent within 30 days of enrollment without approval from the Sponsor/ Investigator (PI). (Off-label use of medication is not considered investigational unless in context of a formal study)
11. History of allergic reaction to 8-MOP
12. Concomitant diagnosis of malignant melanoma or basal cell carcinoma
13. Hypersensitivity or allergy to both heparin and citrate products (if hypersensitive or allergic only to one, exclusion does not apply)
14. Inability to tolerate extracorporeal volume shifts associated with ECP
15. Presence of aphakia
16. History of splenectomy
17. Leucocyte count > 25.000/μl
18. Coagulopathy
19. Known photosensitive disease like systemic lupus erythematosus, porphyrias or albinism

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2020-05-18 (Actual); Primary Completion 2024-06-24 (Actual); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
The proportion of complete response CR (that is, per-cent of patients with skin, liver, and GI GvHD all stage 0) at day 28 of study treatment. | day 28

SECONDARY OUTCOMES:
Overall survival at 1 year | 1 year
Cumulative incidence of NRM | 6 months and at 1 year
Overall response rate (complete response + partial response) | day 28 and day 56
Cumulative incidence of treatment-refractory GvHD | day 28
Cumulative incidence of severe GI GvHD (Grade 3 and 4) | through study completion, an average of 1 year
Time to discontinuation of steroid therapy | Start to end of steroid treatment. Time to discontinuation of steroid treatment will be assessed from start of steroid treatment up to relapse of underlying disease, death from any cause or up to 12 months after start of treatment, whichever came first.
Number of lines of GvHD therapy | through study completion, an average of 1 year
  any additional systemic treatment for GVHD is considered a line of therapy
Cumulative incidence of chronic GvHD | through study completion, an average of 1 year
Number of serious infections | through study completion, an average of 1 year
  defined as grade 3 by the Blood and Marrow Transplant Clinical Trials Network

CONTACTS AND LOCATIONS:
Overall Officials: Francis A. Ayuk, Prof. Dr., Principal Investigator — University Medical Center Hamburg-Eppendorf, Department of Stem Cell Transplantation
Locations (4):
- Medical University of Graz, Department of Internal Medicine, Graz, Austria
- Germany (3):
  - University Medical Center Hamburg-Eppendorf, Hamburg, Hamburg
  - University Hospital Erlangen, Erlangen
  - University Medical Center Regensburg, Regensburg

IPD SHARING:
Plan to Share IPD: No